CLINICAL TRIAL: NCT00857948
Title: A Double-Blind, Placebo-Controlled Study Comparing the Safety and Efficacy of 3 Strengths of Ivermectin Treatment Conditioner and Placebo in Subjects With Pediculus Humanus Capitis (Head Lice) Infestation
Brief Title: Dose Ranging Study of Ivermectin Treatment Conditioner in Subjects With Head Lice Infestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Topaz Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP003
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Pediculus Humanus Capitis (Head Lice)
Keywords: head lice; Pediculus humanus capitis; ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.15% ivermectin (Experimental): Participant on 0.15% ivermectin treatment conditioner
  Interventions: Drug: ivermectin treatment conditioner
- 0.25% ivermectin (Experimental): Participants on 0.25% ivermectin treatment conditioner
  Interventions: Drug: ivermectin treatment conditioner
- 0.50% ivermectin (Experimental): Participants on 0.50% ivermectin treatment conditioner
  Interventions: Drug: ivermectin treatment conditioner
- Placebo (Placebo Comparator): participants on Placebo (Vehicle control)
  Interventions: Drug: Placebo, vehicle control

INTERVENTIONS:
Drug: ivermectin treatment conditioner — Application followed by thorough rinsing of the hair and scalp with water.
  Arms: 0.15% ivermectin; 0.25% ivermectin; 0.50% ivermectin
Drug: Placebo, vehicle control — Application followed by thorough rinsing of the hair and scalp with water.
  Arms: Placebo

SUMMARY:
This is a Phase 2 single center study designed to compare the safety, local tolerability, and efficacy of 3 strengths of ivermectin treatment conditioner to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 6 months old and weighing at least 15 kg.
* Infestation with head lice and viable nits.
* Are otherwise in a normal state of health.
* Willing and able to attend all study visits as scheduled.
* Agree not to cut or chemically treat their hair in the period between treatment and the final visit.
* The subject and/or his/her parent/legal guardian have provided written informed consent, and, if appropriate, the child has provided assent.
* Females of childbearing potential must have a negative urine pregnancy test at screening and agree to take reasonable precautions against becoming pregnant during the study period.

Exclusion Criteria:

* Subjects who have received any over the counter or prescription treatment for head lice in the last 2 weeks.
* Subjects unable to comply with the study obligations and all study visits.
* Subjects with eczema or other chronic conditions of the scalp and skin.
* Subjects in a household with more than 5 infested members.
* Subjects with a history of allergy to ivermectin or any ingredients commonly included in hair products such as shampoos, hair conditioners, or styling aids.
* Subjects with neurologic conditions including a seizure disorder or history of seizures.
* Subjects with an infestation of body lice or pubic lice (determined by questioning).
* Subjects suffering from a condition likely to require medical attention, including administration of oral or systemic antibiotics, oral or systemic corticosteroids, or any other treatment, which in the opinion of the Investigator and visiting physician could influence the results of the study.
* Subjects with other diagnoses which, in the opinion of the Investigator, would interfere with efficacy or safety assessments or would preclude study participation.
* Subjects with very short (shaved) hair.
* Subjects who have been treated with a systemic antibiotic within the previous 2 weeks before screening.
* Subjects who have been previously enrolled in any clinical study within the past 30 days; subjects may not participate in another study while participating in this study.
* Pregnant and/or nursing females.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Topaz
Locations (1):
- Global Health Associates of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Meinking TL, Mertz-Rivera K, Villar ME, Bell M. Assessment of the safety and efficacy of three concentrations of topical ivermectin lotion as a treatment for head lice infestation. Int J Dermatol. 2013 Jan;52(1):106-12. doi: 10.1111/j.1365-4632.2012.05629.x. PMID 23278618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated on 14 March 2009 in 1 US clinical center.
Pre-assignment Details: A total of 78 participants who met the inclusion and exclusion criteria were enrolled and treated.
Groups:
- 0.15% Ivermectin: Participants received a single treatment with 0.15% ivermectin treatment conditioner on Day 1.
- 0.25% Ivermectin: Participants received a single treatment with 0.25% ivermectin treatment conditioner on Day 1.
- 0.50% Ivermectin: Participants received a single treatment with 0.50% ivermectin treatment conditioner on Day 1.
- Placebo: Participants received a single treatment with placebo (treatment conditioner vehicle) on Day 1.
Period: Overall Study
Arm/Group | 0.15% Ivermectin | 0.25% Ivermectin | 0.50% Ivermectin | Placebo
Started | 18 | 18 | 19 | 23
Completed | 15 | 18 | 18 | 23
Not Completed | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.15% Ivermectin | 0.25% Ivermectin | 0.50% Ivermectin | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 19 | 23 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 14 | 13 | 21 | 64
  Between 18 and 65 years | 2 | 4 | 6 | 2 | 14
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 12.28 (13.00) | 14.11 (8.71) | 14.21 (12.87) | 11.13 (8.73) | 12.83 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 18 | 22 | 70
  Male | 3 | 3 | 1 | 1 | 8
Region of Enrollment [Number; unit: Participants]
  United States | 18 | 18 | 19 | 23 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Lice-Free by Day 2 That Were Maintained Through Day 15 Post-treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Live lice eradication was assessed by visual checks of hair and scalp on Days 1, 2 and 8 and by visual checks and counting both live and dead lice from rinse water on Day 15. Eradication was defined as cessation of motility (antennae and leg movement) in all lice.
Time Frame: Day 1 through Day 15 post-application
Population: Live lice eradication was assessed in the Intent-to-treat Population. Any participant with live lice on or after Day 2 received an FDA approved head lice treatment and was classified as a treatment failure, imputed as such for remaining assessments.
Measure: Number; unit: Percent of participants
Arm/Group | 0.15% Ivermectin | 0.25% Ivermectin | 0.50% Ivermectin | Placebo
Number analyzed (Participants) | 18 | 18 | 19 | 23
Percent of participants | 56 | 50 [0 to 0] | 74 [0 to 0] | 9 [0 to 0]

2. Secondary Outcome: Percentage of Index Participants Who Were Lice-Free at Different Time Points Post-treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Live lice eradication was assessed on Days 1, 2, and 8 by visual checks of hair and scalp. Eradication was defined as cessation of motility (antennae and leg movement) in all lice.
Time Frame: Day 1 through Day 8 post-application
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | 0.15% Ivermectin | 0.25% Ivermectin | 0.50% Ivermectin | Placebo
Number analyzed (Participants) | 18 | 18 | 19 | 23
Percent of participants
  Day 1: 2 hours post-application | 33 | 44 [0 to 0] | 32 [0 to 0] | 22 [0 to 0]
  Day 1: 6 hours post-application | 50 | 67 [0 to 0] | 58 [0 to 0] | 30 [0 to 0]
  Day 2 | 83 | 94 [0 to 0] | 95 [0 to 0] | 17 [0 to 0]
  Day 8 | 67 | 72 [0 to 0] | 84 [0 to 0] | 9 [0 to 0]

3. Secondary Outcome: Level of Live Lice Infestation at Different Time Points Post-Treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: The severity of lice infestation was determined by visual checks of hair and scalp. Severity was rated as None: no live lice; Mild: 1 to 5 live lice; Moderate: 6 to 10 live lice; Severe: 11 to 20 live lice; or Very severe > 20 live lice.
Time Frame: Day 1 through Day 15 post-application
Population: The level of lice infestation was assessed in the Intent-to-treat population. Any participant with live lice on or after Day 2 received an FDA approved head lice treatment and was classified as a treatment failure, imputed as such for remaining assessments.
Measure: Number; unit: Percent of participants
Arm/Group | 0.15% Ivermectin | 0.25% Ivermectin | 0.50% Ivermectin | Placebo
Number analyzed (Participants) | 18 | 18 | 19 | 23
Percent of participants
  Day 1: 2 Hours Post Dose: None | 33 | 44 [0 to 0] | 32 [0 to 0] | 22 [0 to 0]
  Day 1: 2 Hours Post Dose: Mild | 50 | 56 [0 to 0] | 63 [0 to 0] | 65 [0 to 0]
  Day 1: 2 Hours Post Dose: Moderate | 17 | 0 [0 to 0] | 5 [0 to 0] | 13 [0 to 0]
  Day 1: 6 Hours Post Dose: None | 50 | 67 [0 to 0] | 58 [0 to 0] | 30 [0 to 0]
  Day 1: 6 Hours Post Dose: Mild | 39 | 33 [0 to 0] | 37 [0 to 0] | 61 [0 to 0]
  Day 1: 6 Hours Post Dose: Moderate | 11 | 0 [0 to 0] | 5 [0 to 0] | 9 [0 to 0]
  Day 2: None | 83 | 94 [0 to 0] | 95 [0 to 0] | 17 [0 to 0]
  Day 2: Mild | 17 | 6 [0 to 0] | 5 [0 to 0] | 78 [0 to 0]
  Day 2: Moderate | 0 | 0 [0 to 0] | 0 [0 to 0] | 4 [0 to 0]
  Day 8: Treatment Failure Day 2 | 17 | 6 [0 to 0] | 5 [0 to 0] | 83 [0 to 0]
  Day 8: None | 72 | 72 [0 to 0] | 84 [0 to 0] | 9 [0 to 0]
  Day 8: Mild | 11 | 6 [0 to 0] | 5 [0 to 0] | 9 [0 to 0]
  Day 8: Moderate | 0 | 6 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Day 8: Severe | 0 | 11 [0 to 0] | 5 [0 to 0] | 0 [0 to 0]
  Day 15: Treatment Failure Day 8 | 33 | 28 [0 to 0] | 16 [0 to 0] | 91 [0 to 0]
  Day 15: None | 56 | 56 [0 to 0] | 74 [0 to 0] | 9 [0 to 0]
  Day 15: Mild | 11 | 17 [0 to 0] | 11 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events Post-treatment With Either Ivermectin or Placebo (Vehicle Control).
Time Frame: Day 1 up to Day 28 post-application
Population: Adverse events were assess in the Safety (Intent-to-treat) Population.
Measure: Number; unit: Participants
Arm/Group | 0.15% Ivermectin | 0.25% Ivermectin | 0.50% Ivermectin | Placebo
Number analyzed (Participants) | 18 | 18 | 19 | 23
Participants
  Conjunctivitis | 0 | 0 [0 to 0] | 1 [0 to 0] | 0 [0 to 0]
  Severe Conjunctivitis | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Eye Pruritus | 1 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Severe Eye Pruritus | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Erythema | 0 | 0 [0 to 0] | 1 [0 to 0] | 3 [0 to 0]
  Severe Erythema | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Folliculitis | 0 | 1 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]
  Severe Folliculitis | 0 | 0 | 0 | 0
  Pruritus | 5 | 1 | 3 | 1
  Severe Pruritus | 0 | 0 | 0 | 0
  Skin Irritation | 0 | 0 | 0 | 1
  Severe Skin Irritation | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 1 up to Day 28 post-application.
Arm/Group | 0.15% Ivermectin | 0.25% Ivermectin | 0.50% Ivermectin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 6/18 | 3/18 | 5/19 | 5/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.15% Ivermectin (N=18) | 0.25% Ivermectin (N=18) | 0.50% Ivermectin (N=19) | Placebo (N=23)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications